CLINICAL TRIAL: NCT01819142
Title: A Multi-Center, Prospective, Cohort Trial Comparing the Effectiveness of AutoloGel Therapy to Usual and Customary Care in Stage II-IV Pressure Ulcers
Brief Title: AutoloGel Therapy to Usual and Customary Care in Pressure Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol study design was re-worked in collaboration with CMS
Sponsor: Cytomedix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM004
Record Dates: First submitted 2013-03-21; First posted 2013-03-27 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Pressure Ulcer
Keywords: non healing wound; pressure ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AutoloGel (Experimental): Subjects will be treated with AutoloGel on average twice a week for the first 2 weeks, and then, once a week thereafter while under active treatment, but actual frequency of treatment will be determined by the treating physician. All patients will receive Autologel treatment
  Interventions: Device: AutoloGel

INTERVENTIONS:
Device: AutoloGel — AutoloGel is a platelet-rich plasma (PRP) gel used in the treatment of non-healing chronic wounds. It will be administered twice weekly for 2 weeks then weekly.
  Other Names: Autologel System

SUMMARY:
The aim of this trial is to demonstrate the effectiveness of complete wound healing in a prospective, open-label, case-matched cohort-controlled trial in which pressure ulcers will be treated using AutoloGel and standard care and case-matched against a concurrent cohort of patients receiving undefined Usual and Customary Care.

DETAILED DESCRIPTION:
Pressure ulcers (PUs) are a common problem in all patient care settings, especially long-term acute care facilities and nursing homes. AutoloGel is a platelet-rich plasma gel used in the treatment of non-healing chronic wounds. The results of AutoloGel to date when used to treat PUs have been promising. The aim of this trial is to demonstrate the effectiveness of complete wound healing in a prospective, open-label, case-matched cohort trial in which pressure ulcers will be treated using AutoloGel and standard of care to determine time to heal at 16 weeks. Comparison will be made with a case matched concurrent cohort of patients receiving undefined Usual and Customary Care.

ELIGIBILITY:
Inclusion Criteria:

1. Medicare/Medicaid eligible
2. ≥18 years of age
3. Ulcer of pressure/shear etiology (Stage II, III, and IV, see Appendix 9 for stage definitions)
4. The largest non-healing wound, if multiple wounds are present, or the single wound to be treated (Index Ulcer) that is located on the heel, ischium, sacrum, and trochanter
5. For subjects with potentially multiple eligible PUs, the largest ulcer will be selected.

   There must be at least 4 cm between the Index Ulcer and other ulcers; if all ulcers are closer than 4 cm, the subject should not be enrolled (screen failure)
6. Debrided ulcer size between 3 cm2 and 200 cm2
7. Demonstrated adequate offloading regimen
8. Duration ≥ 1 month at first visit
9. Subject must be willing to comply with the Protocol, which will be assessed by enrolling clinician.

Exclusion Criteria:

1. Subjects known to be sensitive to AutoloGel components (calcium chloride, thrombin, ascorbic acid) and/or materials of bovine origin
2. Stage I pressure ulcers
3. Ulcers that are unstageable or of deep tissue morphology that have yet to become an open wound
4. Presence of another wound that is concurrently treated and might interfere with treatment of index wound by AutoloGel
5. Ulcer not of PU pathophysiology (e.g., pure diabetic, vasculitic, radiation, rheumatoid, collagen vascular disease, venous, or arterial etiology)
6. Any malignancy other than non-melanoma skin cancer
7. Subjects who are cognitively impaired and do not have a healthcare proxy
8. Serum albumin of less than 2.5 g/dL
9. Plasma Platelet count of less than 100 x 109/L
10. Hemoglobin of less than 10.5 g/dL
11. Subject has inadequate venous access for repeated blood draw required for AutoloGel Administration.

10. Life expectancy of < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Time to complete wound healing | 16 weeks
  Compare complete wound healing at 16 weeks for all pressure ulcers treated with AutoloGel plus standard of care with case-matched concurrent controls. Complete wound closure is defined as skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive study visits 2 weeks apart (FDA Guidance for Industry Chronic Cutaneous Ulcer and Burn Wounds - Developing Products for Treatment, 2006).

SECONDARY OUTCOMES:
Ulcer recurrence | 1 year
  Frequency of ulcer recurrence (recurrence defined as any new ulcer that has appeared since the Index Ulcer healed)
Proportion of healed ulcers | 16 weeks
  Proportion of patients with completely healed pressure ulcers
W-QOL (Quality of Life with Chronic Wounds) score | 16 weeks
  Change in mean W-QOL (Quality of Life with Chronic Wounds) score between baseline and 16 weeks
Number of patients with adverse events as a measure of tolerability | 16 weeks
  Frequency and severity of adverse events during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Singing River, Pascagaula, Mississippi, United States